CLINICAL TRIAL: NCT07124611
Title: Testing the Feasibility of Incorporating Psychosocial Oncology During Neoadjuvant Therapy for Patients With Pancreatic Cancer
Brief Title: A Brief Psychological Intervention to Improve Emotional Well-Being During Neoadjuvant Therapy for Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Jordan Cloyd, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-24234; NCI-2025-05461 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Localized Pancreatic Ductal Adenocarcinoma; Stage 0 Pancreatic Cancer AJCC v8; Stage I Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Interviews as Topic; Nutrition Therapy; Physical Therapy Modalities; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health Services Research (psychosocial care) (Experimental): Patients participate in a psychosocial oncology intervention consisting of meeting with a psychologist via telehealth sessions over 40 minutes once a week for 4 weeks on study. Patients also attend standard physical therapy and nutritional therapy appointments.
  Interventions: Other: Interview; Procedure: Nutritional Therapy; Procedure: Physical Therapy; Behavioral: Psychosocial Care; Other: Questionnaire Administration

INTERVENTIONS:
Other: Interview — Ancillary studies
Procedure: Nutritional Therapy — Attend nutritional appointments
  Other Names: Medical Nutrition Therapy; nutrition therapy
Procedure: Physical Therapy — Attend physical therapy appointments
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
Behavioral: Psychosocial Care — Receive psychosocial care
  Other Names: Psychosocial Support
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well a psychosocial oncology intervention with standard prehabilitation during neoadjuvant therapy works for patients with pancreatic cancer that has not spread to other parts of the body (localized). Chemotherapy and/or radiation therapy prior to surgery, is known as neoadjuvant therapy (NT). The advantages of therapy before surgery include: reducing the size of the cancer mass and/or reducing the spread of cancer, to improve the chance of getting all the cancer during surgery. Other research has shown that doing treatments in this order does lead to improved survival and a lower rate of the cancer returning. Even though there are positives, patients are dealing with emotional and physical symptoms of waiting until the therapies are done to get to surgery. To prepare patients for recovering after chemotherapy and/or radiation therapy to be ready for surgery, care teams have started prehabilitation programs. Prehabilitation includes exercise therapy and nutrition (healthy diet) support before going to surgery. This program has helped boost patients' strength to complete therapies, reduce the number of days in the hospital after surgery and support healing. While meeting with psychologists is available, researchers would like to see if combining it earlier during treatments may provide better support. An oncology (cancer) psychologist while undergoing cancer treatments before surgery may be feasible and helpful to patients with localized pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the feasibility and acceptability of incorporating a psychosocial oncology intervention for patients with pancreatic cancer undergoing neoadjuvant therapy prior to surgical resection.

II. To measure the preliminary efficacy of prehabilitation that includes psychosocial oncology on quality of life and stress/anxiety.

OUTLINE:

Patients participate in a psychosocial oncology intervention consisting of meeting with a psychologist via telehealth sessions over 40 minutes once a week for 4 weeks on study. Patients also attend standard physical therapy and nutritional therapy appointments.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Patient:

  * Newly diagnosed patients with localized pancreatic ductal adenocarcinoma (PDAC) presenting to Ohio State University Wexner Medical Center-Comprehensive Cancer Center (OSUMC-CCC)
  * Plans to initiate neoadjuvant therapy prior to surgical resection
  * Neoadjuvant therapy (NT) and/or surgery may occur at another facility

Exclusion Criteria:

* Prisoners
* Persons unable to provide consent
* Patients unlikely to undergo surgical resection following NT based on anatomical or performance status considerations
* Confirmed or presumed metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the psychosocial oncology intervention | Up to 1 year
  Will be defined as the proportion of enrolled patients who complete the intervention and report that it was acceptable. Will define the incorporation of psychosocial oncology into prehab as feasible and acceptable if >= 70% of enrolled participants agree.

SECONDARY OUTCOMES:
Changes in health-related quality of life for patients with hepatobiliary cancer | Up to 1 year
  Will be assessed using Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep). FACT-Hep consists of the 27-item FACT-G, which assesses generic HRQL concerns, and a validated 18-item Hepatobiliary Subscale (HS), which assesses disease-specific issues. Respondents use a five-point Likert-type scale ranging from 0 to 4, with higher scores reflecting a better quality of life or fewer symptoms. The data will be presented as mean (standard deviation) or median (interquartile range) as appropriate. Differences will be assessed using linear mixed models accounting for within-subject correlations and individual differences.
Changes in mood for patients with hepatobiliary cancer | Up to 1 year
  Will be assessed using the Hospital Anxiety and Depression Scale (HADS). HADS is a 14-item instrument used to measure anxiety and depression in medically ill patients frequently used to identify depression in cancer patients. Scores are totaled for both depression and anxiety symptoms and range from 0 to 21 with a higher score indicating worse symptoms. The data will be presented as mean (standard deviation) or median (interquartile range) as appropriate. Differences will be assessed using linear mixed models accounting for within-subject correlations and individual differences.
Changes in worry for patients with hepatobiliary cancer | Up to 1 year
  Will be assessed using the Penn State Worry Questionnaire (PSWQ). The PSWQ is a 20-item measure of worry. Scores range from 16 to 80 with higher scores indicative of higher levels of worry. The data will be presented as mean (standard deviation) or median (interquartile range) as appropriate. Differences will be assessed using linear mixed models accounting for within-subject correlations and individual differences.
Changes in uncertainty for patients with hepatobiliary cancer | Up to 1 year
  Will be assessed using the Intolerance of Uncertainty Scale (IUS) which Measures a component of worry and anxiety associated with discomfort due to the possibility of future events. Respondents use a five-point Likert-type scale ranging from 1 to 5, with higher scores reflecting a higher intolerance of uncertainty in patients. The data will be presented as mean (standard deviation) or median (interquartile range) as appropriate. Differences will be assessed using linear mixed models accounting for within-subject correlations and individual differences.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan M Cloyd, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu